CLINICAL TRIAL: NCT00448669
Title: Study of the Safety and Efficacy of Daily Oral Antiretroviral Use for the Prevention of HIV Infection in Heterosexually Active Young Adults in Botswana
Brief Title: Botswana TDF/FTC Oral HIV Prophylaxis Trial
Acronym: TDF2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Botswana Ministry of Health (Other Government); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-4940; BOTUSA MB06 (Other: CDC-BOTUSA)
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HIV incidence; HIV prevention; Tenofovir; Emtricitabine; Botswana; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TDF-FTC,condoms,adh/risk counseling (Active Comparator): Eligible participants were randomized to oral Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg (TDF-FTC) once daily in the form of a single tablet. The ratio of randomization was 1:1. Participants randomized to the active arm received male and female condoms, risk reduction counseling, adherence counseling, and routine monitoring for HIV infection, laboratory abnormalities, and adverse events.
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg
- Placebo,condoms,adh/risk counseling (Placebo Comparator): Eligible participants were randomized to the placebo arm and received placebo oral tablets that were visually identical to the TDF-FTC tablet and taken once daily. The placebo tablets contained no active ingredients. The ratio of randomization was 1:1. Participants randomized to the placebo arm received male and female condoms, personalized risk reduction counseling, adherence counseling, and routine monitoring for HIV infection, laboratory abnormalities, and adverse events.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg
  Other Names: Truvada
  Arms: TDF-FTC,condoms,adh/risk counseling
Drug: Placebo Oral Tablet
  Other Names: Placebo
  Arms: Placebo,condoms,adh/risk counseling

SUMMARY:
This study tested whether taking a pill of tenofovir and emtricitabine (two antiretroviral medicines) was safe for sexually-active young adults in Botswana without HIV infection and whether it reduced their risk of getting an HIV infection.

DETAILED DESCRIPTION:
Twelve hundred and nineteen healthy, sexually active women and men, 18-39 years old, without HIV infection were enrolled in Francistown and Gaborone, Botswana. They were provided with free male and female condoms, repeated individualized risk-reduction counseling, diagnosis and treatment of sexually transmitted diseases, and women will be provided with a choice of effective family planning methods. In addition, volunteers were randomized to receive either Tenofovir and emtricitabine (in a single pill) or a placebo pill to take once a day. Volunteers were seen monthly for at least 12 months to monitor for side effects and toxicities and to test their HIV status. Persons who become HIV infected during the trial received ongoing supportive counseling, CD4 and viral load monitoring, education about HIV infection/disease, and access to HIV care including free antiretrovirals when clinically indicated. Volunteer safety was monitored by a local ethics committee, Centers for Disease Control Institutional Review Board (CDC IRB) and an independent data safety and monitoring board

ELIGIBILITY:
Inclusion Criteria:

* citizen of Botswana 18-39 years old
* sexually active
* HIV uninfected
* Hepatitis B and C uninfected
* Calculated creatinine clearance >= 60 mL/min
* hemoglobin >= 8 gm/dL
* ALT and AST <= 2x ULN
* total bilirubin <= 1.5 mg/dL
* total serum amylase <= 1.5x ULN
* Serum phosphorus >= 2.2 mg/dL
* willing to use hormonal contraception (females)
* living within 1 hours travel of study clinic
* pass comprehension test
* willing and able to give informed consent

Exclusion Criteria:

* 18-20 without parent/guardian consent
* history of significant renal or bone disease
* any chronic illness requiring ongoing prescription medication
* pregnant or breastfeeding
* planning to move away from site in the next year
* participating in another HIV prevention or vaccine safety trial
* any other clinical condition or prior therapy that, in the opinion of the study physician, would make the volunteer unsuitable for the study or unable to comply with the dosing requirements

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1219 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Thigpen, MD MPH, Principal Investigator — National Institutes of Health (NIH); Lynn Paxton, MD MPH, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- Centers for Disease Control and Prevention, Atlanta, Georgia, United States
- BOTUSA HIV Prevention Research Unit, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be governed by prevailing CDC data sharing policies.

REFERENCES:
- [Background] Toledo L, McLellan-Lemal E, Henderson FL, Kebaabetswe PM. Knowledge, Attitudes, and Experiences of HIV Pre-Exposure Prophylaxis (PrEP) Trial Participants in Botswana. World J AIDS. 2015 Mar;5(2):10-20. doi: 10.4236/wja.2015.51002. Epub 2015 Feb 12. PMID 26767149
- [Background] Kasonde M, Niska RW, Rose C, Henderson FL, Segolodi TM, Turner K, Smith DK, Thigpen MC, Paxton LA. Bone mineral density changes among HIV-uninfected young adults in a randomised trial of pre-exposure prophylaxis with tenofovir-emtricitabine or placebo in Botswana. PLoS One. 2014 Mar 13;9(3):e90111. doi: 10.1371/journal.pone.0090111. eCollection 2014. PMID 24625530
- [Background] Chirwa LI, Johnson JA, Niska RW, Segolodi TM, Henderson FL, Rose CE, Li JF, Thigpen MC, Matlhaba O, Paxton LA, Brooks JT. CD4(+) cell count, viral load, and drug resistance patterns among heterosexual breakthrough HIV infections in a study of oral preexposure prophylaxis. AIDS. 2014 Jan 14;28(2):223-6. doi: 10.1097/QAD.0000000000000102. PMID 24361682
- [Background] Kebaabetswe PM, Stirratt MJ, McLellan-Lemal E, Henderson FL, Gray SC, Rose CE, Williams T, Paxton LA. Factors Associated with Adherence and Concordance Between Measurement Strategies in an HIV Daily Oral Tenofovir/Emtricitibine as Pre-exposure Prophylaxis (Prep) Clinical Trial, Botswana, 2007-2010. AIDS Behav. 2015 May;19(5):758-69. doi: 10.1007/s10461-014-0891-z. PMID 25186785
- [Background] Segolodi TM, Henderson FL, Rose CE, Turner KT, Zeh C, Fonjungo PN, Niska R, Hart C, Paxton LA. Normal laboratory reference intervals among healthy adults screened for a HIV pre-exposure prophylaxis clinical trial in Botswana. PLoS One. 2014 Apr 8;9(4):e93034. doi: 10.1371/journal.pone.0093034. eCollection 2014. PMID 24714095
- [Result] Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT; TDF2 Study Group. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med. 2012 Aug 2;367(5):423-34. doi: 10.1056/NEJMoa1110711. Epub 2012 Jul 11. PMID 22784038
- [Result] Gust DA, Soud F, Hardnett FP, Malotte CK, Rose C, Kebaabetswe P, Makgekgenene L, Henderson F, Paxton L, Segolodi T, Kilmarx PH. Evaluation of Sexual Risk Behavior Among Study Participants in the TDF2 PrEP Study Among Heterosexual Adults in Botswana. J Acquir Immune Defic Syndr. 2016 Dec 15;73(5):556-563. doi: 10.1097/QAI.0000000000001143. PMID 27509251

RESULTS

PARTICIPANT FLOW:
Groups:
- TDF-FTC, Condoms, Risk Counseling: Participants randomized to the active arm received daily oral TDF-FTC along with male and female condoms, personalized risk reduction counseling, adherence counseling, and routine monitoring for HIV infection, laboratory abnormalities, and adverse events.
  Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg: Daily oral single dose pill containing 300 mg TDF and 200 mg FTC.
- Placebo, Condoms, Risk Counseling: Participants randomized to the placebo arm received a daily oral placebo tablet along with male and female condoms, personalized risk reduction counseling, adherence counseling, and routine monitoring for HIV infection, laboratory abnormalities, and adverse events.
  TDF-FTC placebo: Placebo comparator for TDF-FTC
Period: Overall Study
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Started | 611 | 608
Completed | 393 | 410
Not Completed | 218 | 198
Not completed — Lost to Follow-up | 52 | 63
Not completed — Withdrawal by Subject | 90 | 74
Not completed — Relocated | 49 | 36
Not completed — Were withdrawn by investigator | 10 | 6
Not completed — Death | 2 | 4
Not completed — Had other reasons | 5 | 6
Not completed — HIV-infected at enrollment | 1 | 2
Not completed — Never started drug | 9 | 7

BASELINE CHARACTERISTICS:
Population: A total of 1219 underwent randomization. Of the 611 assigned to TDF-FTC: 9 did not start TDF-FTC and 1 was HIV-infected at enrollment. Of the 608 assigned to placebo: 7 did not start placebo and 2 were HIV-infected at enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling | Total
Number analyzed (Participants) | 611 | 608 | 1219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 611 | 608 | 1219
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 277 | 557
  Male | 331 | 331 | 662
Region of Enrollment [Number; unit: participants]
  Botswana | 611 | 608 | 1219

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions in the Tenofovir/Emtricitabine and Placebo Arms
Description: Study visits were scheduled every 30 days until completion of the study, and participants were instructed to return to the clinic for evaluation in the event of an illness. Participants reported any adverse effects at monthly visits and interim visits.
Time Frame: Monthly, for up to 3 years
Measure: Number; unit: percentage of participants with AE
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Number analyzed (Participants) | 611 | 608
percentage of participants with AE | 91.2 | 88.2
Statistical Analysis 1: Comparison: TDF-FTC, Condoms, Risk Counseling vs Placebo, Condoms, Risk Counseling; Safety analyses were performed in the intention-to-treat cohort. Primary safety end points included the frequency of adverse clinical or laboratory events; Test type: Superiority or Other; p = 0.003, Regression, Cox

2. Primary Outcome: HIV Incidence in the Tenofovir/Emtricitabine and Placebo Arms
Description: Study visits were scheduled every 30 days until completion of the study and during monthly study visits, we performed testing for HIV infection. At completion of the study, we tested all participants for HIV infection, using an enzyme-linked immunosorbent assay (ELISA).The primary efficacy end point was the difference in the rates of HIV infection between participants assigned to receive TDF-FTC and those assigned to receive placebo. The initial efficacy analysis included all study participants who were randomly assigned to receive a study medication (intention-to-treat cohort).
Time Frame: Monthly, for up to 3 years
Population: Of the 1219, 3 were excluded from analysis because HIV-infected at the time of enrollment.
Measure: Number; unit: infections/100 person-years
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Number analyzed (Participants) | 610 | 606
infections/100 person-years | 1.2 | 3.1
Statistical Analysis 1: Comparison: TDF-FTC, Condoms, Risk Counseling vs Placebo, Condoms, Risk Counseling; The primary efficacy end point was the difference in the rates of HIV infection between participants assigned to receive TDF-FTC and those assigned to receive placebo. The primary hypothesis was that TDF-FTC, as compared with placebo, would reduce the rate of HIV infection by at least 65%, with a predefined lower boundary for the 95% confidence interval of 10%; Test type: Superiority or Other; p = 0.03, Regression, Cox; Efficacy = 62.2, 95% CI 2-sided [21.5 to 83.4]

3. Secondary Outcome: Changes in Condom Use During Study: Number of Participants With >=1 Condomless Sex Acts
Description: We assessed condom use of the enrolled participants by face-to-face interviews (at baseline and monthly thereafter) and provided a comprehensive package of HIV prevention services, including individualized counseling on risk reduction, free male and female condoms, and screening for sexually transmitted infections followed, if applicable, by partner notification and treatment.
Time Frame: 12 months
Population: Of 1219, 19 excluded (3 HIV-infected at enrollment, 16 never started drug). Of the 1200, 24 reported no sex during study. Remaining total 1176 with >=1 sex act included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Number analyzed (Participants) | 611 | 608
Participants
  Baseline: number analyzed (Participants) | 506 | 503
  Baseline | 124 | 113
  Month 1: number analyzed (Participants) | 449 | 441
  Month 1 | 94 | 86
  Month 2: number analyzed (Participants) | 414 | 410
  Month 2 | 97 | 90
  Month 3: number analyzed (Participants) | 376 | 358
  Month 3 | 92 | 83
  Month 4: number analyzed (Participants) | 357 | 326
  Month 4 | 73 | 66
  Month 5: number analyzed (Participants) | 339 | 326
  Month 5 | 67 | 61
  Month 6: number analyzed (Participants) | 323 | 341
  Month 6 | 70 | 67
  Month 7: number analyzed (Participants) | 293 | 292
  Month 7 | 55 | 45
  Month 8: number analyzed (Participants) | 255 | 266
  Month 8 | 57 | 49
  Month 9: number analyzed (Participants) | 240 | 243
  Month 9 | 55 | 45
  Month 10: number analyzed (Participants) | 209 | 214
  Month 10 | 51 | 36
  Month 11: number analyzed (Participants) | 195 | 201
  Month 11 | 36 | 33
  Month 12: number analyzed (Participants) | 185 | 195
  Month 12 | 54 | 30
Statistical Analysis 1: Comparison: TDF-FTC, Condoms, Risk Counseling; A logistic regression was used to estimate the odds of reporting zero condomless sex acts. The longitudinal dependent variable (number of condomless sex acts) was defined as: Number of condomless vaginal sexual acts with both casual and main partners among those who reported having had at least one sexual partner in the previous 30 days; Test type: Superiority or Other; p = 0.004, Regression, Logistic; In this univariate model with the analysis of number of condomless sex acts, our model estimates the odds of reporting no condomless sex acts; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.05 to 1.28]

4. Secondary Outcome: Rates of Adherence to Study Medication
Description: The rates of adherence to study medication by treatment arm was assessed over the entire course of the study. This comparison was done by assessing the percentage of pills taken by participants within each study arm. The difference between the 2 arms was compared with a Fisher' exact test.
Time Frame: 36 months
Measure: Mean (Standard Deviation); unit: Percentage of pills taken
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Number analyzed (Participants) | 611 | 608
Percentage of pills taken | 93.5 (0.136) | 93.6 (0.137)
Statistical Analysis 1: Comparison: TDF-FTC, Condoms, Risk Counseling vs Placebo, Condoms, Risk Counseling; Fisher's Exact Test was performed to test for differences between the treatment groups in terms of adherence based on pill count; Test type: Superiority or Other; p = 0.79, Fisher Exact

5. Secondary Outcome: Antiretroviral (ARV) Resistance Patterns in Seroconverters
Description: Participants who seroconverted had blood samples taken at the time of infection and at one month and six months post seroconversion to detect any HIV resistance mutations.
Time Frame: At time HIV infection diagnosed,1 month post-time of HIV infection diagnosis, and 6 months post-time of HIV infection diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Number analyzed (Participants) | 10 | 26
Participants | 1 | 1

6. Secondary Outcome: CD4 Evaluation After HIV Seroconversion
Description: Study medication was stopped when HIV infected was diagnosed. Seroconvertors were referred for clinical care and followed an additional year with scheduled quarterly CD4+ cell count assessments. A model-estimated geometric mean of the CD4+ cell counts by each treatment group was evaluated.
Time Frame: 1-year post seroconversion
Measure: Geometric Mean (95% Confidence Interval); unit: cells/microliter
Groups:
- TDF-FTC Seroconvertor Group: Participants who were assigned to receive TDF-FTC and seroconverted.
- Placebo Seroconvertor Group: Participants who were assigned to receive the placebo and seroconverted.
Arm/Group | TDF-FTC Seroconvertor Group | Placebo Seroconvertor Group
Number analyzed (Participants) | 9 | 24
cells/microliter | 500 [378 to 661] | 466 [396 to 549]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the course of the study until study completion, i.e. up to 3 years.
Description: Adverse events were graded according to the National Institutes of Health Division of AIDS (DAIDS) Table for Grading Severity of Adult and Pediatric Adverse Events (December 2004).
Arm/Group | TDF-FTC, Condoms, Risk Counseling | Placebo, Condoms, Risk Counseling
Serious Adverse Events (participants affected / at risk) | 42/611 | 44/608
Other Adverse Events (participants affected / at risk) | 557/611 | 536/608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF-FTC, Condoms, Risk Counseling (N=611) | Placebo, Condoms, Risk Counseling (N=608)
Elevated ALT (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperamylasemia (Endocrine disorders) | 9 (11) | 9 (18)
Hyperchloremia (General disorders) | 1 (1) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Renal and urinary disorders) | 20 (21) | 21 (24)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypernatremia (Renal and urinary disorders) | 1 (1) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Headache (General disorders) | 2 (2) | 1 (1)
Injury, non-fatal (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tonsillitis, acute (Infections and infestations) | 1 (1) | 1 (1)
Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF-FTC, Condoms, Risk Counseling (N=611) | Placebo, Condoms, Risk Counseling (N=608)
Abnormal Menses (Reproductive system and breast disorders) | 54 (68) | 64 (79)
Abscess (Skin and subcutaneous tissue disorders) | 13 (13) | 17 (18)
Acne (Skin and subcutaneous tissue disorders) | 11 (11) | 5 (5)
Allergy, unspecified (General disorders) | 9 (9) | 6 (6)
Anorexia (Gastrointestinal disorders) | 17 (17) | 15 (16)
Balanitis (Reproductive system and breast disorders) | 6 (6) | 8 (11)
Bite (Injury, poisoning and procedural complications) | 5 (6) | 10 (11)
Breast Abnormalities (Reproductive system and breast disorders) | 7 (7) | 10 (10)
Chest Pain (Cardiac disorders) | 28 (34) | 39 (44)
Chlamydia (Reproductive system and breast disorders) | 76 (85) | 75 (83)
Upper Respiratory Infection (Infections and infestations) | 231 (385) | 241 (439)
Conjuctivitis (Eye disorders) | 20 (20) | 20 (22)
Constipation (Gastrointestinal disorders) | 29 (33) | 23 (24)
Contusion (Skin and subcutaneous tissue disorders) | 8 (10) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (36) | 39 (44)
Dermatitis (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7)
Dermatomycosis (Skin and subcutaneous tissue disorders) | 14 (14) | 5 (6)
Dermatophytosis (Skin and subcutaneous tissue disorders) | 34 (35) | 24 (26)
Diarrhea (Gastrointestinal disorders) | 76 (93) | 65 (76)
Disturbance of Skin Sensation (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (3)
Dizziness (Nervous system disorders) | 92 (109) | 65 (80)
Dysmenorrhea (Reproductive system and breast disorders) | 32 (47) | 34 (46)
Dysuria (Renal and urinary disorders) | 17 (24) | 24 (29)
Edema, limb (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (8)
Epistaxis (General disorders) | 6 (7) | 8 (8)
Fatigue (General disorders) | 53 (55) | 45 (48)
Fever (General disorders) | 11 (11) | 11 (11)
Flatulence (Gastrointestinal disorders) | 56 (67) | 58 (63)
Folliculitis (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (10)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Gastroesophageal Reflux (Gastrointestinal disorders) | 9 (12) | 4 (4)
Generalized Pain (General disorders) | 11 (11) | 6 (6)
Genital Herpes (Reproductive system and breast disorders) | 28 (43) | 35 (46)
Gonorrhea (Reproductive system and breast disorders) | 28 (32) | 18 (21)
Headache (General disorders) | 225 (384) | 225 (410)
Hypertension (Cardiac disorders) | 6 (6) | 13 (13)
Hypotension (Cardiac disorders) | 7 (7) | 3 (3)
Injury, Nonfatal (Injury, poisoning and procedural complications) | 13 (13) | 15 (18)
Leukorrhea (Reproductive system and breast disorders) | 30 (39) | 53 (64)
Myalgia (Musculoskeletal and connective tissue disorders) | 17 (19) | 23 (25)
Nausea (Gastrointestinal disorders) | 113 (132) | 43 (48)
Oral Disease, Gingiva (General disorders) | 10 (11) | 4 (4)
Oral Disease, Teeth (General disorders) | 33 (43) | 40 (51)
Pain, Ear (Ear and labyrinth disorders) | 3 (3) | 10 (10)
Pain, Abdominal (Gastrointestinal disorders) | 154 (214) | 156 (217)
Pain, Acute Musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (8)
Pain, Back (Musculoskeletal and connective tissue disorders) | 57 (72) | 67 (89)
Pain, Genital (Reproductive system and breast disorders) | 7 (8) | 8 (9)
Pain, Joint (Musculoskeletal and connective tissue disorders) | 28 (34) | 23 (27)
Pain, Limb (Musculoskeletal and connective tissue disorders) | 21 (24) | 28 (31)
Painful Eyes (Eye disorders) | 7 (8) | 8 (9)
Palpitations (Cardiac disorders) | 18 (21) | 15 (20)
Pelvic Inflammatory Disease (Reproductive system and breast disorders) | 7 (9) | 11 (12)
Pharyngitis, Acute (General disorders) | 39 (45) | 37 (38)
Polyphagia (Endocrine disorders) | 35 (38) | 30 (33)
Pruritus, Genital (Reproductive system and breast disorders) | 15 (16) | 19 (20)
Pruritus, Unspecified (Skin and subcutaneous tissue disorders) | 12 (12) | 12 (12)
Rash, Unspecified (Skin and subcutaneous tissue disorders) | 39 (44) | 42 (48)
Rhinitis (General disorders) | 6 (7) | 7 (7)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 12 (14)
Sore Ulcer, Genital (Reproductive system and breast disorders) | 12 (12) | 6 (7)
Sore Ulcer, Oral Cavity (Skin and subcutaneous tissue disorders) | 9 (11) | 5 (5)
Tonsilitis, Acute (General disorders) | 24 (28) | 24 (24)
Trichomoniasis (Reproductive system and breast disorders) | 20 (21) | 18 (23)
Urethral Discharge (Reproductive system and breast disorders) | 2 (2) | 11 (15)
Urinary Tract Infection (Renal and urinary disorders) | 8 (10) | 9 (9)
Vaginal Candidiasis (Reproductive system and breast disorders) | 38 (42) | 28 (37)
Vomiting (Gastrointestinal disorders) | 69 (87) | 43 (47)
Wound (Skin and subcutaneous tissue disorders) | 33 (37) | 34 (40)
Blood Urea Nitrogen (Renal and urinary disorders) | 2 (2) | 1 (1)
Phosphate (Blood and lymphatic system disorders) | 122 (198) | 138 (221)
Amylase, Serum (Gastrointestinal disorders) | 306 (986) | 293 (999)
AST/SGOT (Gastrointestinal disorders) | 36 (43) | 38 (42)
ALT/SGPT (Gastrointestinal disorders) | 37 (47) | 43 (66)
Bilirubin, total (Blood and lymphatic system disorders) | 41 (70) | 39 (73)
Bilirubin, direct (Gastrointestinal disorders) | 17 (19) | 17 (25)
Sodium (Blood and lymphatic system disorders) | 126 (172) | 113 (148)
Potassium (Blood and lymphatic system disorders) | 24 (27) | 22 (25)
Bicarbonate (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Chloride (Blood and lymphatic system disorders) | 25 (30) | 21 (23)

LIMITATIONS AND CAVEATS:
The rates of study completion were lower than predicted because more participants withdrew from the study, mostly due to relocation or conflicting obligations.Findings may not be generalizable to other populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No